CLINICAL TRIAL: NCT02006953
Title: Bolus Versus Continuous Feeding Regimens Post Gastrostomy Tube Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting due to parent declining feeding strategy
Sponsor: University of Michigan (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Steven W. Bruch, M.D., MSc., Clinical Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00046483
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Enteral Nutrition; Enteral Feeding; Gastrostomy Tube
Keywords: gastrostomy; enteral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus (Active Comparator): Bolus: Total volume of feedings is determined by the amount of formula required to meet calorie and protein needs, which is determined by a Registered Dietitian. Volume of each bolus is determined by dividing the total volume of feeding by the desired number of feedings per day:
  If child is less than 6 months: 8 feeds/day If child is 6-12 months 6 feeds/day If child is 12 months or greater: 5 feedings/day Rate of feeds is determine by the rate needed to infuse each bolus over 1 hour. Patient to remain NPO. Once at goal, if able to take PO, may offer orally first with remainder of goal volume over the remainder of the hour.
  Interventions: Procedure: Bolus feeding schedule following gastrostomy tube placement
- Continuous (Active Comparator): Continuous: Total volume of feedings is determined by the amount of formula required to meet calorie and protein needs, which is determined by a Registered Dietitian. Rate of feeds is determined by dividing total volume of feedings by 24 hours. Patient is to remain NPO. Once at goal, if able to take PO, may offer hourly amount orally, but only 2x per day.
  Interventions: Procedure: Continuous chimney feeds following gastrostomy tube placement

INTERVENTIONS:
Procedure: Bolus feeding schedule following gastrostomy tube placement
  Arms: Bolus
Procedure: Continuous chimney feeds following gastrostomy tube placement
  Arms: Continuous

SUMMARY:
The purpose of this study is to determine the best way to feed children after they have a gastrostomy tube placed. The study compares bolus feeding to continuous feeding.

DETAILED DESCRIPTION:
This study will consist of a prospective, randomized comparison of bolus versus continuous enteral feeding protocols in pediatric patients with gastrostomy tubes

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age
* Admitted for gastrostomy tube placement, with or without Nissen Fundoplication

Exclusion Criteria:

* Immunocompromised patients
* Short Bowel Syndrome (SBS)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2011-08; Primary Completion 2018-07-18 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Rate of gastrostomy tube leakage | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.

SECONDARY OUTCOMES:
Emesis | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.
Retching | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.
Venting beyond recommendations | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.
Feeding changes | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.
Unscheduled clinic/ER visits/calls | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.
G-tube infection | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.
Weight | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.
Time to goal feeds | 8 weeks
  Symptoms are rated by parents on a daily diary for the first 4 weeks following g-tube placement, and then on a weekly diary for the next 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Bruch, MD, MSc, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, CS Mott Children's Hospital, Ann Arbor, Michigan
  - Mercy Children's Hospital, Toledo, Ohio